CLINICAL TRIAL: NCT01768481
Title: Intervention précoce Sur Les Indices d'athérogénèse Des Adolescents à Risque
Brief Title: Intima Media Thickness Regression in Dyslipidemic Teenagers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Laurent Legault, associate professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMR
Record Dates: First submitted 2013-01-08; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Obesity; Dyslipidemia
Keywords: Obesity; Dyslipidemia; Cholesterol; Intima media thickness
MeSH Terms: conditions — Obesity; Dyslipidemias | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Statin (Experimental): Atorvastatin 10 mg every day for one year
  Interventions: Drug: Atorvastatin
- Sugar pill (Placebo Comparator): Same size, taste and size placebo tablet (manufactured by sponsor) given every day for one year.
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Atorvastatin — 10 mg Atorvastatin vs placebo daily in a randomized controlled trial for one year
  Other Names: Statin; Lipitor
  Arms: Statin
Drug: sugar pill — placebo controlled arm receives similarly looking placebo.
  Other Names: placebo
  Arms: Sugar pill

SUMMARY:
Randomized controlled trial of statin intervention in dyslipidemic obese teenagers. Primary outcome is intima media thickness before and after intervention.

DETAILED DESCRIPTION:
Obese teenagers with abnormal lipid profiles were randomized to either low dose statin or placebo and had their carotid intima media thickness compared before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Obesity
* Abnormal Triglyceride levels (>1.7mmol/L).
* Abnormal HDL-C levels (1.0mmol/L)

Exclusion Criteria:

* Abnormal thyroid unfction (not treated)
* Diabetes

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2004-01; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
carotid intima media thickness | 12 months
  Carotid Intima media thickness measured at baseline and after 12 months in 2 arms (placebo and statin)

SECONDARY OUTCOMES:
weight | 12 months
  weight, height and BMI recorded before and after intervention

OTHER OUTCOMES:
Lipid profile | 6 months
  Complete lipid profile were recorded at baseline , 6 months and 12 months after intervention.
lipid profile | 12 months
  Lipid profile measured at end of study
BMI | 12 months
  BMI neasured at baseline and at end of study
liver functions | 3 months
  ALT/AST done at 3, 6, 9 and 12 months
liver functions | 6 months
  ALT/AST done at 3, 6, 9, and 12 months
liver functions | 9 months
  ALT/AST done at 3, 6, 9, and 12 months
liver functions | 12 months
  ALT/AST done at 3, 6, 9, and 12 months
creatinine kinase | 3 months
  CK done at 3 , 6, 9 and 12 months
creatinine kinase | 6 months
  CK done at 3 , 6, 9 and 12 months
creatinine kinase | 9 months
  CK done at 3 , 6, 9 and 12 months
creatinine kinase | 12 months
  CK done at 3 , 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Legault, MD, Principal Investigator — Hopital Maisonneuve-Rosemont, UMontreal
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada